CLINICAL TRIAL: NCT04914611
Title: Real World Assessment of People Living With Chronic Hepatitis B in Australia
Acronym: REACH-B
Status: Recruiting | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHCRP2008
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBsAg Positive: Patients with chronic hepatitis B infection as defined by HBV surface antigen positive
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The REACH-B study establishes an observational cohort study of people living with chronic hepatitis B from a national network, including a diverse range of services, to characterise and monitor hepatitis B linkage to care and treatment requirements amongst this population.

DETAILED DESCRIPTION:
Participants presenting to participating clinics for HBV care within the previous 12 months will be identified and enrolment data will be collected including demographics, laboratory parameters, liver disease assessment, treatment history and clinical management. Follow-up data on HBV treatment and clinical management, liver disease stage and laboratory parameters will be collected at each subsequent visit or at minimum every 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals diagnosed with chronic hepatitis B in the participating study sites are eligible to be included (both newly diagnosed cases and those diagnosed in the past).
2. 16 years of age or older.
3. Attended the health service for HBV care within the prior 12 months from study commencement (retrospective recruitment) OR Attending the health service for HBV care from study commencement (prospective recruitment)

Exclusion Criteria:

1. Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with chronic HBV as defined by a positive HBsAg result at participating sites will be enrolled in the cohort. Participants can be newly diagnosed or existing patients of the service. Data on HBV disease status, liver disease status, HBV monitoring and treatment will be collected six monthly from enrolment.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Characterisation of HBV | July 2027
  To characterise and monitor hepatitis B linkage to care and treatment requirements amongst people living with chronic hepatitis B

SECONDARY OUTCOMES:
Socio-demographics of HBV infected population | July 2027
  To characterise the socio-demographic spectrum of people living with chronic HBV
HBV Disease staging | July 2027
  To assess the proportion of individuals in each phase of the disease, based on the natural history of hepatitis B infection
HBV Care Cascade | July 2027
  To assess the proportion of individuals who are eligible for each recommended hepatitis B clinical care level
HBV Treatment and Care | July 2027
  To monitor the uptake of recommended hepatitis B clinical care, including antiviral treatment
HBV Care and treatment adherence | July 2027
  To monitor the adherence to recommended hepatitis B care, including the patterns of antiviral use and cessation
HCC Surveillance | July 2027
  To assess the rate of surveillance for hepatocellular carcinoma
HBV Disease Progression | July 2027
  To assess the rate of progression from each phase to the subsequent phase of hepatitis B
Liver fibrosis progression | July 2027
  To assess the rate of liver fibrosis progression, including the development of cirrhosis, decompensated cirrhosis, and hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, PhD MBBS, Principal Investigator — Kirby Insitute, UNSW
Locations (19):
- Australia (19):
  - Australasian Society for HIV, Viral Hepatitis and Sexual Health Medicine (ASHM), Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Justice Health and Forensic Mental Health Network, Sydney, New South Wales
  - Blacktown Mount Druitt Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Menzies School of Health Research (Royal Darwin & Alice Springs Hospitals), Darwin, Northern Territory
  - Top End Medical Centre, Darwin, Northern Territory
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Cairns and Hinterland Hospital Health Service, Cairns, Queensland
  - Torres and Cape Hospital and Health Service, Cairns, Queensland
  - Central Adelaide Local Health Network (Royal Adelaide & The Queen Elizabeth Hospitals), Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Cohealth, Melbourne, Victoria
  - Utopia Refugee and Asylum Seeker Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Albany Health Campus, WACHS Great Southern, Albany, Western Australia
  - Broome Regional Hospital, WACHS Kimberley, Broome, Western Australia
  - Kalgoorlie Health Campus, WACHS Goldfields, Kalgoorlie-Boulder, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided